CLINICAL TRIAL: NCT06150651
Title: Safety/Phase I Study of PiggyBac Transposon Mediated Chimeric Antigen Receptor T Cells Targeting CD-19 in Thai Patients With Refractory Systemic Lupus Erythematosus
Brief Title: Safety of PiggyBac Transposon CAR T-cells Targeting CD-19 in Refractory Lupus.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other); Health Systems Research Institute,Thailand (Other Government)
Responsible Party: Principal Investigator, Wonngarm Kittanamongkolchai, MD, Principle Investigator, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLE-PB-CD19-CART
Record Dates: First submitted 2023-11-13; First posted 2023-11-29 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: SLE (Systemic Lupus)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: Intervention: PiggyBac transposon-mediated CD-19 CAR T-cells (1x10^6 cells/kg)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR T-cell therapy (Experimental): Subjects will receive a conditioning lymphodepletion chemotherapy regimen of fludarabine and cyclophosphamide, followed by the infusion of 1x10^6 cells/kg CD-19 CAR-T cells.
  Interventions: Other: CAR T-cell therapy

INTERVENTIONS:
Other: CAR T-cell therapy — 1x10^6 cells/kg CD-19 CAR-T cells

SUMMARY:
A Phase 1 clinical trial to evaluate the safety and efficacy of PiggyBac transposon-mediated Chimeric Antigen Receptor(CAR) T-cells targeting CD19 in refractory Systemic Lupus Erythematosus (SLE) patients who have not responded to standard immunosuppressive treatments.

DETAILED DESCRIPTION:
This is a single-institution phase I study in adults with refractory SLE. Autologous Peripheral Blood Mononuclear Cells will be transduced with a chimeric antigen receptor targeting the B-cell surface antigen CD19 using the PiggyBac Transposon system. Subjects will receive a conditioning lymphodepletion chemotherapy regimen of fludarabine and cyclophosphamide, followed by the infusion of 1x10^6 cells/kg CD-19 CAR T-cells. Subjects will be evaluated post-treatment for toxicity, SLE disease activity, and the persistence of CAR-expressing T cells in vivo.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years.
2. Diagnosis of Systemic Lupus Erythematosus (SLE), as defined by the American College of Rheumatology (ACR) 1997 criteria, The Systemic Lupus International Collaborating Clinics (SLICC) criteria, or the European Alliance of Associations for Rheumatology (EULAR)/ACR classification.
3. Refractory SLE, defined by one or more of the following:

   3.1 Persistently active SLE requiring ongoing maintenance therapy (if not contraindicated) with:
   * Antimalarial drug.
   * Either mycophenolate (minimum daily dose of 1500 mg) or azathioprine (minimum daily dose of 1.5 mg/kg).
   * Patients must also need a minimum daily dose of 7.5 mg prednisolone for lower disease activity maintenance, or have a SLEDAI score of 8 or higher.

   3.2 Biopsy-proven proliferative lupus nephritis after two standard induction therapies, including intravenous cyclophosphamide (cumulative dose of at least 1.5 g) and mycophenolate mofetil (administered for a minimum of 3 months), unless contraindicated.

   3.3 Worsening of biopsy-proven lupus nephritis (activity index > 6 and chronicity index < 6 within 6 months), indicated by increased proteinuria and/or decreased estimated glomerular filtration rate, despite treatment with high-dose corticosteroids (prednisolone at least 0.7 mg/kg/day or equivalent) and either mycophenolate mofetil or cyclophosphamide for a minimum of 14 days.
4. Ability to understand and willingness to sign a written informed consent document.
5. Participants of child-bearing or child-fathering potential must agree to practice birth control from enrollment until four months after receiving CAR T-cell infusion.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. History of active malignancy, excluding non-melanoma skin cancer and carcinoma in situ (e.g., cervix, bladder, breast).
3. History of vital organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities, cirrhosis, or psychiatric illness/social situations that limit compliance with study requirements.
5. Any other clinically significant disease history or current disease that, in the judgment of the research physician, may pose a risk to the safety of the subjects or interfere with the research procedure, or the evaluation of safety and efficacy.
6. Serologic status indicating active HIV, hepatitis B, or C infection. Participants positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative PCR prior to enrollment.
7. History of severe adverse drug reaction to Cyclophosphamide or Fludarabine.
8. Received a live vaccine within 30 days prior to CAR-T cell infusion.
9. eGFR CKD-EPI < 30 ml/min/1.73m^2.
10. Participation in other clinical investigations during the study period.
11. Prior receipt of CAR-T cell therapy outside this protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety of PiggyBac transposon-mediated CAR T-cell infusion targeting CD19 in adult patients with refractory SLE. | Up to 28 days after CD-19 CAR-T cell infusion
  The incidence of adverse events assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0

SECONDARY OUTCOMES:
Disease activity of SLE | 3, 6, and 12 months after CD-19 CAR-T cell infusion
  The Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA) - Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)
Complete response rate of lupus nephritis | 3, 6, and 12 months after CD-19 CAR-T cell infusion
  Complete response defined as normal or ≤ 25% decline of estimated glomerular filtration rate (eGFR) Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) from baseline and urinary protein to creatinine index (UPCI) or 24-hour urinary protein ≤ 0.5 g/g or g/day
Partial response rate of lupus nephritis | 3, 6, and 12 months after CD-19 CAR-T cell infusion
  Partial response defined as normal or ≤25% decline of eGFR CKD-EPI from baseline and at least 50% reduction of proteinuria, with a UPCI or 24-hour urinary protein between 0.5 to 3 g/g or g/day

CONTACTS AND LOCATIONS:
Overall Officials: Wonngarm Kittanamongkolchai, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Please Select, Thailand

IPD SHARING:
Plan to Share IPD: No